CLINICAL TRIAL: NCT04937660
Title: Palbociclib Combinations in HR+/HER2- Metastatic Breast Cancer Patients: A Non-Interventional Prospective Study on the Treatment Patterns & Clinical Outcomes in Africa Middle East (PRECIOUS)
Brief Title: Treatment Patterns & Clinical Outcomes of Palbociclib Combinations in HR+HER2-MBC
Acronym: PRECIOUS
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A5481150; PRECIOUS (Other: Alias Study Number)
Record Dates: First submitted 2021-06-08; First posted 2021-06-24 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Metastatic Breast Cancer
Keywords: Palbociclib; Africa; Middle East
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of this non-interventional multicenter study is to provide prospective, observational data on patients initiating treatment with palbociclib combination to contribute to the knowledge of HR+ HER2-metastatic/locally advanced Breast Cancer (BC) disease management, its treatment pattern, clinical outcomes and quality of life (QoL) in the routine clinical practice in Africa and Middle East countries .

DETAILED DESCRIPTION:
Patients with HR+/HER2- metastatic/locally advanced BC whose treatment decision with palbociclib has been made by their treating physician and who meet the eligibility criteria will be invited to participate in the study. Patients who initiate treatment with palbociclib plus letrozole/aromatase inhibitor or palbociclib plus fulvestrant in line with the licensed indication(s), as first or second line therapy for metastatic/locally advanced BC at enrollment may be included in the study.

The variables assessed in this study will be patient demographics, clinical characteristics, comorbid conditions and concomitant medications, HR+ HER2-locally advanced and metastatic BC treatment history, current BC treatment, performance status (Eastern Cooperative Oncology Group (ECOG), clinical outcomes, and QoL. All assessments described in this protocol are performed as part of normal clinical practice or standard practice guidelines for the patient population and healthcare provider specialty in the countries where this non-interventional study is being conducted. All data collected in this study are intended to capture the real-world treatment patterns and outcomes for patients with HR+/HER2- metastatic/locally advanced BC. An electronic case report form (eCRF) will be used for data collection. Investigators will be trained with an initial on-site visit to the clinic on the protocol, electronic data capture (EDC) system (i.e., eCRF), investigator site master file (ISMF), documentation, and any applicable study processes. Any new information relevant to the performance of this non-interventional study (NIS) will be forwarded to the medical staff during the study. Remote data monitoring will be conducted during the life of the study to ensure timely reporting of safety data, data integrity and consistency.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years or older with diagnosis of adenocarcinoma of the breast with evidence of metastatic /locally advanced disease not amenable to treatment with curative intent.
2. Documented HR+ (ER+ and/or PR+) tumor based on local standards
3. Documented HER2- tumor based on local standards
4. Will initiate treatment with palbociclib plus letrozole/aromatase inhibitor or palbociclib plus fulvestrant in line with the licensed indication(s), as first or second line therapy for metastatic/locally advanced BC at enrollment
5. Patients who in the opinion of the investigator are willing and able to comply with regular clinic visits
6. Evidence of a personally signed and dated informed consent document indicating that the patient (or a legally acceptable representative) has been informed of all pertinent aspects of the study

Exclusion Criteria:

1. Patients participating in any interventional clinical trial
2. Patients on active treatment for malignancies other than metastatic/locally advanced BC at the time of enrollment
3. Patients who are unable to understand the nature of the study and are unwilling to sign an informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with HR+/HER2- metastatic/locally advanced Breast Cancer
Sampling Method: Non-Probability Sample
Enrollment: 185 (Actual)
Dates: Start 2021-07-15 (Actual); Primary Completion 2025-04-29 (Actual); Study Completion 2025-04-29 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival | Baseline up to 24 months
  The period from study entry until disease progression, or death
Overall Survival | Baseline up to 24 months
  Overall Survival is defined as the time from the date of start of palbociclib combination treatment till the date of death due to any cause.

SECONDARY OUTCOMES:
Objective Response Rate | 2 years
  Tumor response to treatment; Complete response, partial response, or stable disease

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (12):
- Egypt (4):
  - Alexandria School of Medicine/Clinical Research Center CRC, Alexandria
  - Dar El Salam Oncology Hospital, Cairo
  - National Cancer Institute, Cairo
  - Ain Shams University Hospital, Cairo
- King Hussein Cancer Center, Amman, Jordan
- Lebanon (4):
  - American University of Beirut Medical Center, Beirut
  - Hôtel Dieu de France (HDF), Beirut
  - Saint Joseph Hospital - Cancer Centers of Colorado, Jdeidé - Metn
  - Hammoud Hospital University Medical Center (HHUMC), Sidon
- Hamad Medical Corporation, Doha, Qatar
- Saudi Arabia (2):
  - King Fahad Specialist Hospital KFSH-Dammam, Dammam
  - National Guard Hospital, Riyadh, Riyadh

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A5481150